CLINICAL TRIAL: NCT02549716
Title: Clinical, Pharmacological and Molecular Effects of Intravenous and Oral Acetaminophen in Adults With Aneurysmal Sub-Arachnoid Hemorrhage
Brief Title: Clinical, Pharmacological and Molecular Effects of IV and Oral Acetaminophen in Adults With aSAH
Acronym: aSAH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding was stopped
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sprague W Hazard III, Assistant Professor of Anesthesiology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRBSTUDY00002767
Record Dates: First submitted 2015-07-01; First posted 2015-09-15 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Subarachnoid Hemorrhage; Stroke
Keywords: Acetaminophen; interleukin-6; interleukin-1; thromboxane A2
MeSH Terms: conditions — Subarachnoid Hemorrhage; Stroke | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV acetaminophen + oral placebo (Experimental): Patients in this group will receive IV acetaminophen and an oral placebo. The IV formulation will be given using the FDA approved OFIRMEV which comes in a single glass bottle at a concentration of 1000mg/100ml (10mg/ml) containing a total of 1 gram of acetaminophen.
  Interventions: Drug: IV acetaminophen; Drug: Oral placebo
- Oral acetaminophen + IV placebo (Experimental): Patients in this group will receive oral acetaminophen and a saline solution placebo through their IV. The enteral formulation will be in the standard tablet form of 500mg per pill. Patients will receive two pills, or 1 gram of acetaminophen.
  Interventions: Drug: Oral acetaminophen; Drug: IV placebo

INTERVENTIONS:
Drug: IV acetaminophen — Patients in this group will receive IV acetaminophen and an oral placebo every 6 hours for a 14 day period. Blood and CSF samples will be collected from patients throughout the 14 day period.
  Other Names: Ofirmev; IV paracetamol
  Arms: IV acetaminophen + oral placebo
Drug: Oral acetaminophen — Patients in this group will receive oral acetaminophen and an IV saline solution placebo every 6 hours for a 14 day period. Blood and CSF samples will be collected from patients throughout the 14 day period.
  Other Names: Tylenol; paracetamol
  Arms: Oral acetaminophen + IV placebo
Drug: Oral placebo — Patients who receive IV acetaminophen will also receive an oral placebo with their IV treatments (every 6 hours for a 14 day period).
  Other Names: placebo
  Arms: IV acetaminophen + oral placebo
Drug: IV placebo — Patients who receive oral acetaminophen will also receive a saline solution placebo at the same time that they receive the oral acetaminophen treatment (every 6 hours for 14 days).
  Other Names: placebo, saline solution
  Arms: Oral acetaminophen + IV placebo

SUMMARY:
This study compares the bioavailability of IV and PO acetaminophen in both blood and the cerebrospinal fluid (CSF) of patients following subarachnoid hemorrhage. The study will also compare the temperature and levels of inflammatory cytokines in both blood and CSF of patients treated with IV and PO acetaminophen.

DETAILED DESCRIPTION:
In individuals diagnosed with subarachnoid hemorrhage (SAH), fevers have been shown to have detrimental micro and macroscopic effects on the brain that can ultimately cause secondary brain injury. The anti-pyretic effects of oral acetaminophen have been studied in critically ill patients but no study has been able to compare these effects to the IV form of acetaminophen also known as OFIRMEV. The investigators wish to explore the notion that IV acetaminophen will be more effective than enteral acetaminophen in reducing the incidence of non-infectious fevers in critically ill patients. In addition, the investigators propose to study the levels of inflammatory cytokines after administration of IV or enteral acetaminophen, as well as, determine the incidence of vasospasm in SAH patients treated with IV acetaminophen. Currently, external ventricular drain (EVD) placement is the "standard of care" in patients who present with SAH and altered mental status/coma. The presence of an EVD allows for continuous sampling and removal of cerebral spinal fluid (CSF) as necessary to alleviate dangerous elevations in intracranial pressure. This clinical scenario allows for a unique, continuous outlet to access the CSF, without placing patients at risk, and without further invasive procedures (i.e. repeated spinal taps). These samples of CSF can be assayed for levels of acetaminophen, as well as inflammatory markers of fever which include interleukin-1 (IL-1), interleukin-6 (IL-6), and thromboxane-2 (TXA-2), in patients selected to be given enteral or IV acetaminophen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subarachnoid hemorrhage (must be confirmed by CT, CT angiography, lumbar puncture, or MRI).
* Fisher Grade between 1-3 (subarachnoid blood without signs of intraventricular hemorrhage or parenchymal extension).
* Placement of an external ventricular drain.
* Adults aged 18-100 years.

Exclusion Criteria:

* Anyone under the age of 18 or over the age of 100.
* Adult patients with subarachnoid hemorrhage with interventricular hemorrhage or parenchymal extension (Fisher Grade 4).
* Contraindication to acetaminophen such as a known hypersensitivity, severe hepatic impairment, or severe active liver disease.
* Severe renal impairment (creatinine clearance ≤ 30 mL/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sprague W Hazard, MD, Principal Investigator — "Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Acetaminophen + Oral Placebo | Oral Acetaminophen + IV Placebo
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen + Oral Placebo | Oral Acetaminophen + IV Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 37 [37 to 37] | 45 [45 to 46] | 42.6 [37 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Bioavailability of Acetaminophen in Cerebral Spinal Fluid (CSF) and Blood
Description: Patients in both IV and PO groups will have samples taken from their Cerebral Spinal Fluid (CSF) and blood at the above times after acetaminophen is administered for the first time. They will then have additional samples taken every 24 hours following the time of first drug administration for 14 days. Patients will also have a sample collected every 35 hours (1 hour before the 6th loading dose) to determine the steady state level of acetaminophen.
Time Frame: Time = 0, 5, 15, 30, 45, 60, 90, 120, 180, 240, and 360 minutes after first drug administration
Population: Outcome measure was not analyzed because study was terminated early.
Arm/Group | IV Acetaminophen + Oral Placebo | Oral Acetaminophen + IV Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Concentrations of Interleukin-1 (IL-1), Interleukin-6 (IL-6), and Thromboxane A-2 (TXA-2) in Cerebral Spinal Fluid (CSF) and Blood
Description: Patients in both IV and PO groups will have samples taken from their Cerebral Spinal Fluid (CSF) and blood at the above times after acetaminophen is administered for the first time. They will then have additional samples taken every 24 hours following the time of first drug administration for 14 days. These samples will be examined to determine concentrations of Interleukin-1 (IL-1), Interleukin-6 (IL-6), and thromboxane A-2 (TXA-2) in both the Cerebral Spinal Fluid (CSF) and blood. This will enable the team to determine if route of entry of acetaminophen plays a significant role in the level of inflammatory markers in critically ill patients.
Time Frame: Time = 0, 5, 15, 30, 45, 60, 90, 120, 180, 240, and 360 minutes after first drug administration. Additionally, every 24 hours after time t=0 for 14 days (14 additional samples from both blood and CSF).
Population: Outcome measure was not analyzed because study was terminated early
Arm/Group | IV Acetaminophen + Oral Placebo | Oral Acetaminophen + IV Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Febrile Periods
Description: Patients in both IV and PO groups will have their temperatures taken at the times listed. This will help determine if route of entry of acetaminophen plays a significant role in the number of febrile periods.
Time Frame: as for outcome 2
Population: Outcome measure was not analyzed because study was terminated early
Arm/Group | IV Acetaminophen + Oral Placebo | Oral Acetaminophen + IV Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Incidence of Vasospasm
Description: The investigators will measure the incidence of vasospasm in patients with subarachnoid hemorrhage (SAH) who receive 1g Q6 of IV acetaminophen starting on post-bleed day 0 and continuing for 14 consecutive days (typical vasospasm window). Clinical vasospasm will be defined as the presence of new focal neurological deficits (motor or speech deficits) that developed after subarachnoid hemorrhage (SAH), a decrease in the Glasgow Coma Score (GCS) of 2 or more points for >6hrs, a new cerebral infarction unrelated to post-treatment (coiling or clipping) complications, re-bleed, progressive hydrocephalus, electrolyte or metabolic disturbance, or infection. The incidence of clinical vasospasm will be identified in the patients Electronic Medical Record (EMR) after the 14 day period.
Time Frame: Days 0-14 following diagnosis with subarachnoid hemorrhage.
Population: Outcome measure was not analyzed because study was terminated early.
Arm/Group | IV Acetaminophen + Oral Placebo | Oral Acetaminophen + IV Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks (14 days)
Arm/Group | IV Acetaminophen + Oral Placebo | Oral Acetaminophen + IV Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Acetaminophen + Oral Placebo (N=1) | Oral Acetaminophen + IV Placebo (N=2)
Elevated Liver Function Tests (Hepatobiliary disorders) | 0 (0) | 1 (1) — A participant was had an elevation in liver function tests that were greater than three times the admission values and led to withdrawal from the study

LIMITATIONS AND CAVEATS:
Study was terminated early

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT02549716/Prot_SAP_000.pdf